CLINICAL TRIAL: NCT02637726
Title: Bispectral Index Under Propofol Anesthesia in Children : a Comparative Randomised Study Between TIVA and TCI
Brief Title: Bispectral Index Under Propofol Anesthesia in Children : a Study Between TIVA and TCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pr Isabelle CONSTANT (Other)
Responsible Party: Sponsor-Investigator, Pr Isabelle CONSTANT, Professor Isabelle Constant, Hôpital Armand Trousseau
Organization: Hôpital Armand Trousseau (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIVCM
Record Dates: First submitted 2015-12-16; First posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Anesthesia
Keywords: Total intravenous anesthesia; Target Controlled Infusion; Propofol; Bispectral index; Children
MeSH Terms: interventions — Consciousness Monitors; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- TIVA0 (Experimental): Propofol : TIVA guided by clinical signs. Remifentanil
  Interventions: Drug: Propofol : TIVA; Drug: Remifentanil
- TIVA BIS (Experimental): propofol : TIVA guided by EEG Monitoring. Remifentanil
  Interventions: Drug: Propofol : TIVA; Device: EEG Monitoring; Drug: Remifentanil
- TCI KBIS (Experimental): Propofol : TCI Kataria guided by EEG Monitoring. Remifentanil.
  Interventions: Drug: Propofol : TCI Kataria; Device: EEG Monitoring; Drug: Remifentanil
- TCI SBIS (Experimental): Propofol : TCI Schnider guided by EEG Monitoring. Remifentanil.
  Interventions: Drug: Propofol : TCI Schnider; Device: EEG Monitoring; Drug: Remifentanil

INTERVENTIONS:
Drug: Propofol : TCI Schnider — Target controlled infusion using schnider model for propofol
  Arms: TCI SBIS
Drug: Propofol : TCI Kataria — Target controlled infusion using Kataria model for propofol
  Arms: TCI KBIS
Drug: Propofol : TIVA — Total intravenous anesthesia without use of a pharmokinetic model
  Arms: TIVA BIS; TIVA0
Device: EEG Monitoring — Maintaining a bispectral index between 45 and 55
  Other Names: BISPECTRAL INDEX
  Arms: TCI KBIS; TCI SBIS; TIVA BIS
Drug: Remifentanil — Remifentanil at discretion of the anesthesiologist

SUMMARY:
In children, only a few studies have compared different modes of propofol infusion during a total intravenous anesthesia (TIVA) with propofol and remifentanil. The aim of this study is to compare Bispectral Index (BIS) profiles (percentage of time spent at adequate BIS values) between four modes of propofol infusion: titration of the infusion rate on clinical signs (TIVA0), titration of the infusion rate on the BIS (TIVABIS), target controlled infusion (TCI) guided by the BIS either with the Kataria model (TCI KBIS) or the Schnider model (TCI SBIS).

Methods: Children will be prospectively randomized into the 4 groups. In the TIVA0 group the anesthesiologist is blinded to the BIS. In each group, the percentage of time with adequate BIS values (45-55), the bias and imprecision will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* weighting more than 15 kg;
* American Society of Anesthesiologists physical status I or II
* scheduled for middle ear surgery

Exclusion Criteria:

* cardiovascular, neurological, hepatic or renal impairment, if their body mass index was above 95th percentile or if they received any drug interfering with the central nervous system.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2006-02; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Percentage of time spent at adequate BIS values | from the beginning to the end of the anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Constant, PhD, Study Director — Hôpital Armand Trousseau
Locations (1):
- Departement d'anesthesie Hopital Armand Trousseau, Paris, France

IPD SHARING:
Plan to Share IPD: No